CLINICAL TRIAL: NCT01050023
Title: Provant Therapy of Venous Stasis Ulcer Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southern California Institute for Research and Education (Other)
Collaborators: Regenesis Biomedical, Inc. (Industry)
Responsible Party: Ian Gordon, M.D., Ph.D., VA Long Beach Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #965
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Venous Stasis Ulcers
Keywords: venous stasis ulcer; wound healing; Provant Wound Closure System; radiofrequency; Provant; pain relief
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 - Active Treatment (Experimental): Provant device activated to emit RF energy
  Interventions: Device: Provant Device (Wound Therapy System)
- 2 - Inactive Treatment (Sham Comparator): Provant device not activated to emit RF energy
  Interventions: Device: Provant Device - Inactive

INTERVENTIONS:
Device: Provant Device (Wound Therapy System) — Twice daily application of the active Provant device to the wound for twelve (12) weeks.
  Arms: 1 - Active Treatment
Device: Provant Device - Inactive — Twice daily application of the inactive Provant device to the wound for twelve (12) weeks.
  Arms: 2 - Inactive Treatment

SUMMARY:
This pilot study hypothesizes that use of the Regenesis Provant Wound Therapy System (a radiofrequency device) twice daily over venous stasis ulcers (wounds thought to occur due to improper functioning of valves in the veins, usually of the legs) will result in increased rates of healing and a larger proportion of completely healed wounds after 12 weeks of therapy compared to wounds treated identically using a Provant device that is not activated to emit radiofrequency.

ELIGIBILITY:
Inclusion Criteria:

* Ulcer size between 1.0 and 16.0 cm2 at the time of randomization - measurements to be taken after sharp debridement if this is performed at the screening visit. Wounds must be free of necrotic tissue and fibrin slough after debridement with at least 90% of the surface covered with granulation tissue.
* Target ulcer must be present for at least 6 weeks prior to randomization. Other ulcers close to the study ulcer are allowable and may be any size but should be greater than 2cm away from the study ulcer; no more than 4 ulcers total on the target limb are allowed.
* A duplex ultrasound study documenting venous disease must be performed within on year of study entry. The ultrasound exam should document either chronic occlusion of the target limb popliteal, femoral, or iliac veins or the vena cava, or occlusion in the greater or lesser saphenous veins, or reflux in either the deep, saphenous, or perforating veins.

Exclusion Criteria:

* No ulcer on the target limb including the study ulcer may be deep enough to expose structures deep to the adipose lay of skin such as muscle, fascia, tendon, joint, or bone. The presence of sinus tracts that have not been sufficiently marsupialized such that the wound depth can be assessed by gross visual inspection is similarly exclusion.
* At the Screening or Randomization Visits, the presence of significant periwound cellulitis or the need to administer systemic antibiotics. system antibiotic therapy for any indication within 10 days of screening is an exclusion.
* Baseline arterial studies obtained within one year of screening or at the screening visit must show either an ankle-brachial index of the affected limb greater or equal to 0.75 based on the higher of the two pedal arteries systolic pressure measured with Doppler ultrasound compared to the ipsilateral brachial artery systolic pressure determined with Doppler ultrasound.
* Any major surgery or trauma affecting the target limb such as tibial fracture, knee arthroplasty, endovascular or open arterial or venous surgery or femoral stenting within 180 days of randomization.
* Participation in any clinical trial involving therapy for wound healing within 30 days of randomization.
* Concurrent administration of systemic agents that influence wound healing such as prednisone or dexamethasone in any quantity, cytotoxic chemotherapy agents, or immunosuppressive therapy.
* Previous ionizing radiation therapy at any dose near the wound bed (within 5 cm).
* A history of cancer in the target limb except for previous skin cancer treated in the target limb provided that a biopsy of the target wound is obtained within 90 days of randomization that confirms the absence of neoplasia.
* Severe renal failure - serum creatinine greater than 2.5 or subject on hemodialysis.
* Severe hepatic insufficiency: known cirrhosis, any degree of ascites, serum transamines more than three times the upper limit of normal.
* Known allergy or intolerance to cadexomeric iodine or latex free Profore bandages.
* The presence of 1) implanted pacemaker, automatic defibrillator, neurostimulator, bone stimulators, cochlear implants, or other devices with metal leads; 2) implanted or programmable pumps or intravenous or intrathecal drug delivery; 3) metal implant within 25 cm of area of treatment.
* Pregnancy. Women of childbearing potential must agree to use adequate contraception.
* Live expectancy of last than one year.
* Uncompensated or uncontrolled right heart failure with associated edema.
* Inability to walk independently (adaptive devices such as walkers or canes are allowed).
* BMI greater than 50.
* Severe anemia, hemoglobin less than 8.5
* Poorly controlled diabetes, A1cHgb greater than 12
* Severe hypoalbuminemia, serum albumen less than 2.6.
* Active local or systemic malignancy such as lung cancer or leukemia
* Severe hypertension - systolic bp greater than 180 or diastolic bp greater than 100
* Severe hypoxemia - chronic oxygen or ventilator therapy.
* HIV infection unless on retroviral therapy and viral load undetectable by PCR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Rates of wound closure (measured as change in surface area - mm2/day) | during and after 12 weeks of therapy

SECONDARY OUTCOMES:
Proportion of wounds achieving complete healing | afer 12 weeks of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ian Gordon, M.D., Ph.D., Principal Investigator — VA Long Beach Healthcare System
Locations (2):
- United States (2):
  - VA Long Beach Healthcare System, Long Beach, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California